CLINICAL TRIAL: NCT07352436
Title: Prospective Cohort Study on the Impact of Gut Microbiota and Serum Metabolites on Glycemic Variability and Clinical Outcomes in Patients With Diabetic Kidney Disease
Brief Title: Gut Microbiota and Serum Metabolites as Predictors of Glycemic Variability and Outcomes in Diabetic Kidney Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Eighth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: PY-2025-04
Record Dates: First submitted 2025-11-24; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetic Kidney Disease; Glycemic Variability; Gut Microbiota
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples，Stool samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetic kidney disease (DKD) is one of the main complications of diabetes and a leading cause of end-stage kidney disease. Blood glucose variability is closely associated with disease progression in individuals with DKD. Recent evidence suggests that gut bacteria and their circulating metabolites may play important roles in regulating blood glucose variability and clinical outcomes. However, it remains unclear whether gut bacteria and blood metabolites influence DKD progression through effects on blood glucose variability.

This study aims to (1) characterize gut bacteria and blood metabolites in individuals with DKD at different stages and levels of disease severity, and evaluate their value in predicting adverse outcomes; (2) assess the relationships among gut bacteria, blood metabolites, and blood glucose variability; and (3) determine whether gut bacteria and blood metabolites affect clinical outcomes by modulating blood glucose variability.

A total of 270 individuals with DKD will be enrolled in a prospective observational cohort. The investigators will conduct continuous glucose monitoring and collect stool and blood samples for advanced analyses of gut microbiota and blood metabolites. The objective is to clarify how gut bacteria and circulating metabolites relate to blood glucose variability and disease prognosis, and to develop tools to identify high-risk individuals at an early stage. Ultimately, the findings may provide new insights and strategies to improve clinical care and quality of life for individuals with DKD.

DETAILED DESCRIPTION:
Diabetic kidney disease (DKD) is a major microvascular complication of diabetes and a leading cause of end-stage kidney disease. Blood glucose variability (GV) has been shown to be closely associated with disease progression in individuals with DKD. Recent studies suggest that gut microbiota and their serum metabolites may play important roles in regulating GV and influencing clinical outcomes. However, it remains unclear whether gut microbiota and serum metabolites affect DKD progression through GV.

This prospective observational cohort study aims to address three key questions:

1. Characterize gut microbiota and serum metabolites in individuals with DKD at different disease stages and severities, and evaluate their prognostic value for adverse outcomes.
2. Examine the relationships among gut microbiota, serum metabolites, and blood glucose variability.
3. Determine whether gut microbiota and serum metabolites influence clinical outcomes by affecting blood glucose variability.
4. A total of 270 individuals with DKD will be enrolled. The investigators will conduct continuous glucose monitoring (CGM), collect blood and stool samples, and analyze these samples using 16S rRNA high-throughput sequencing and untargeted serum LC-MS. These data will be used to assess GV, characterize gut microbiota and serum metabolites, and develop predictive models for adverse outcomes in DKD. The study aims to clarify the impact of gut microbiota and blood glucose variability on DKD prognosis and to develop tools for early identification of high-risk individuals, ultimately improving disease management and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Diagnosis of Diabetic Kidney Disease (DKD)
3. Type 2 Diabetes Mellitus
4. Stable Antidiabetic Regimen:The antidiabetic regimen must have been stable for at least 3 months prior to study enrollment.
5. Willingness to Provide Informed Consent:

Participants must voluntarily sign an informed consent form to participate in the study. -

Exclusion Criteria:

1. Acute Diabetic Complications:

   Participants with acute diabetic complications, such as diabetic ketoacidosis (DKA), or with primary kidney diseases like primary glomerulonephritis, nephrotic syndrome, or lupus nephritis.
2. Infection or Stress Conditions:

   Participants in a state of infection, trauma, or other stress conditions.
3. Pregnancy or Lactation:

   Women who are pregnant, breastfeeding, or planning to become pregnant in the next month.
4. Severe Dermatologic Conditions:

   Participants with severe dermatologic conditions, such as extensive eczema, widespread scars, tattoos, herpetic dermatitis, severe edema, or psoriasis.
5. Skin Issues with Sensor Application:

   Participants with severe skin issues at the site of sensor application, such as burns, injuries, sunburns, ulcers, or scars from prior surgery.
6. Coagulation or Blood Disorders:

   Participants with abnormal coagulation, anemia, or abnormal hematocrit.
7. Chronic Gastrointestinal Diseases or Surgery History:

   Participants with chronic gastrointestinal diseases or a history of gastrointestinal or biliary surgery.
8. Recent Probiotic or Antibiotic Use:

Participants who have used probiotics or prebiotics, or received antibiotic treatment for more than 3 days in the past 3 months, or have consumed yogurt or yogurt-containing foods/beverages in the past week.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients diagnosed with Diabetic Kidney Disease (DKD), aged between 18 and 65 years. All participants will have a confirmed diagnosis of Type 2 Diabetes Mellitus (T2DM) in accordance with the 1999 World Health Organization diagnostic criteria, and meet the diagnostic criteria for DKD as outlined in the 2021 Chinese Guidelines for the Prevention and Treatment of Diabetic Kidney Disease.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Diabetic Kidney Disease (DKD) Progression | Time Frame: 12 months (from baseline to endpoint assessment) This time frame reflects the follow-up period during which DKD progression will be monitored in the study cohort.
  DKD progression is defined as the occurrence of at least one of the following events: (1) end-stage kidney disease requiring dialysis or kidney transplantation; or (2) a sustained decline of ≥30% in estimated glomerular filtration rate (eGFR) from baseline. This outcome will be used to assess the predictive value of blood glucose variability, gut microbiota, serum metabolites, and inflammatory markers for long-term DKD progression.

SECONDARY OUTCOMES:
Number of Participants with Cardiovascular Mortality | Time Frame: 12 months Adverse events will be monitored over a period of 12 months from baseline to track occurrences and assess their relationship with GV and other biomarkers.
  Cardiovascular mortality is defined as death resulting from heart disease or related cardiovascular complications occurring during the follow-up period.
Number of Participants with Major Adverse Cardiovascular Events (MACE) | 12 months (from baseline)
  Major adverse cardiovascular events (MACE) are defined as the occurrence of myocardial infarction, stroke, or unstable angina during the follow-up period.
Number of Participants Undergoing Kidney Transplantation | 12 months (from baseline)
  Kidney transplantation is defined as receipt of a kidney transplant procedure during the follow-up period.
Number of Participants with Hypoglycemic Events | 12 months (from baseline)
  Hypoglycemic events are defined as documented episodes of hypoglycemia occurring during the study period, identified by continuous glucose monitoring and/or clinical records.

DOCUMENTS (2):
  • Study Protocol (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT07352436/Prot_000.pdf
  • Informed Consent Form (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT07352436/ICF_001.pdf